CLINICAL TRIAL: NCT07294911
Title: Predictors of Contrast-Induced Acute Kidney Injury in Patients With Acute Coronary Syndrome
Brief Title: Predictors of Contrast-induced Acute Renal Injury in Patients With Acute Coronary Syndrome
Acronym: PC-AKI-ACS
Status: Completed | Type: Observational
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CI-AKI-STEMI-2025
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndrome; Contrast-Induced Acute Kidney Injury
Keywords: Contrast-induced nephropathy; Contrast-induced acute kidney injury; Acute coronary syndrome; Percutaneous coronary intervention; STEMI; NSTEMI; Risk factors; Predictors; Renal dysfunction; CI-AKI
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples collected after contrast exposure are stored at -80°C for the analysis of biomarkers of kidney injury, including TIMP-2. No DNA will be extracted or analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Coronary Syndrome Patients Undergoing PCI: Patients admitted with acute coronary syndrome (STEMI or NSTEMI) who underwent coronary angiography or percutaneous coronary intervention. Clinical, laboratory, and procedural data were collected to identify predictors of contrast-induced acute kidney injury (CI-AKI). No additional interventions were applied beyond standard clinical care.
  Interventions: Other: Observational data collection

INTERVENTIONS:
Other: Observational data collection — Data collected from routine clinical care to evaluate predictors of contrast-induced acute kidney injury after PCI. No intervention applied.

SUMMARY:
This observational study aims to identify predictors of contrast-induced acute kidney injury (CI-AKI) in patients with acute coronary syndrome undergoing percutaneous coronary intervention. Clinical, laboratory, and procedural factors will be analyzed to determine their association with the development of CI-AKI. The findings may help improve risk stratification and preventive strategies in this high-risk population.

DETAILED DESCRIPTION:
This prospective observational study investigates predictors of contrast-induced acute kidney injury (CI-AKI) among patients with acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI). The study was conducted from November 2024 to June 2025 at a tertiary cardiac center.

Patients with ACS who underwent coronary angiography or PCI were enrolled consecutively. Clinical characteristics, laboratory parameters, hydration status, use of nephrotoxic drugs, and type and volume of contrast media were recorded. Serum creatinine levels were measured before and 48-72 hours after contrast exposure, and CI-AKI was defined according to KDIGO criteria.

The primary objective is to identify independent predictors of CI-AKI using multivariate analysis. Secondary objectives include evaluation of short-term outcomes, such as in-hospital complications and renal function recovery at 90 days. The results are expected to improve understanding of CI-AKI risk in real-world ACS patients and to support preventive strategies in interventional cardiology.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Diagnosis of acute coronary syndrome (STEMI or NSTEMI) confirmed by clinical, ECG, and laboratory findings

Undergoing coronary angiography or percutaneous coronary intervention with intravascular contrast administration

Provided informed consent to participate in the study

Availability of baseline and follow-up serum creatinine values

Exclusion Criteria:

Known chronic kidney disease stage 4 or 5 (eGFR < 30 mL/min/1.73 m²) or on dialysis

Hemodynamic instability not related to acute coronary syndrome (e.g., septic shock)

Exposure to intravenous contrast within the previous 7 days

Use of nephrotoxic drugs (e.g., aminoglycosides, amphotericin B) within 72 hours prior to contrast exposure

Active infection or inflammatory disease affecting renal function

Pregnancy or breastfeeding

Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years old) with ST-segment elevation myocardial infarction (STEMI) who underwent emergency percutaneous coronary intervention with intravascular contrast. Participants were prospectively enrolled between November 2024 and June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Change in serum creatinine at 90 days | 90 days after contrast exposure
  Change in serum creatinine level compared to baseline at 90-day follow-up after contrast exposure, to evaluate renal function recovery or persistent impairment.
Incidence of Contrast-Induced Acute Kidney Injury (CI-AKI) | Within 72 hours after contrast exposure
  Occurrence of contrast-induced acute kidney injury (CI-AKI) defined as an increase in serum creatinine of ≥0.3 mg/dL (≥26.5 µmol/L) or ≥50% from baseline within 48-72 hours after exposure to iodinated contrast media, according to KDIGO criteria.

SECONDARY OUTCOMES:
Changes in plasma TIMP-2 concentration | 2 hours after contrast exposure
  Assessment of urinary TIMP-2 levels 2 hours after contrast exposure to detect early markers of renal tubular injury

CONTACTS AND LOCATIONS:
Overall Officials: Miras M Mugazov, MD, PhD, Principal Investigator — Karaganda Medical University
Locations (1):
- Karaganda Medical University, Karaganda, Qaraghandy Oblysy, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and institutional policy restrictions. Aggregate results may be available upon reasonable request after publication.

REFERENCES:
- [Background] Koyner JL, Shaw AD, Chawla LS, Hoste EA, Bihorac A, Kashani K, Haase M, Shi J, Kellum JA; Sapphire Investigators. Tissue Inhibitor Metalloproteinase-2 (TIMP-2)⋅IGF-Binding Protein-7 (IGFBP7) Levels Are Associated with Adverse Long-Term Outcomes in Patients with AKI. J Am Soc Nephrol. 2015 Jul;26(7):1747-54. doi: 10.1681/ASN.2014060556. Epub 2014 Dec 22. PMID 25535301
- [Background] Martin-Cleary C, Sanz AB, Avello A, Sanchez-Nino MD, Ortiz A. NephroCheck at 10: addressing unmet needs in AKI diagnosis and risk stratification. Clin Kidney J. 2023 Jun 22;16(9):1359-1366. doi: 10.1093/ckj/sfad146. eCollection 2023 Sep. PMID 37664563
- [Background] Ortega LM, Heung M. The use of cell cycle arrest biomarkers in the early detection of acute kidney injury. Is this the new renal troponin? Nefrologia (Engl Ed). 2018 Jul-Aug;38(4):361-367. doi: 10.1016/j.nefro.2017.11.013. Epub 2018 Apr 5. English, Spanish. PMID 29627229
- [Background] Sun Q, Kang Z, Li Z, Xun M. Urinary NGAL, IGFBP-7, and TIMP-2: novel biomarkers to predict contrast medium-induced acute kidney injury in children. Ren Fail. 2022 Dec;44(1):1201-1206. doi: 10.1080/0886022X.2022.2075277. PMID 36120960
- [Background] Gonzalez-Nicolas MA, Gonzalez-Guerrero C, Goicoechea M, Bosca L, Valino-Rivas L, Lazaro A. Biomarkers in Contrast-Induced Acute Kidney Injury: Towards A New Perspective. Int J Mol Sci. 2024 Mar 19;25(6):3438. doi: 10.3390/ijms25063438. PMID 38542410
- [Background] Fahling M, Seeliger E, Patzak A, Persson PB. Understanding and preventing contrast-induced acute kidney injury. Nat Rev Nephrol. 2017 Mar;13(3):169-180. doi: 10.1038/nrneph.2016.196. Epub 2017 Jan 31. PMID 28138128
- [Background] McDonald JS, McDonald RJ, Carter RE, Katzberg RW, Kallmes DF, Williamson EE. Risk of intravenous contrast material-mediated acute kidney injury: a propensity score-matched study stratified by baseline-estimated glomerular filtration rate. Radiology. 2014 Apr;271(1):65-73. doi: 10.1148/radiol.13130775. Epub 2014 Jan 16. PMID 24475854
- [Background] McDonald RJ, McDonald JS, Carter RE, Hartman RP, Katzberg RW, Kallmes DF, Williamson EE. Intravenous contrast material exposure is not an independent risk factor for dialysis or mortality. Radiology. 2014 Dec;273(3):714-25. doi: 10.1148/radiol.14132418. Epub 2014 Sep 9. PMID 25203000
- [Background] Hinson JS, Ehmann MR, Fine DM, Fishman EK, Toerper MF, Rothman RE, Klein EY. Risk of Acute Kidney Injury After Intravenous Contrast Media Administration. Ann Emerg Med. 2017 May;69(5):577-586.e4. doi: 10.1016/j.annemergmed.2016.11.021. Epub 2017 Jan 25. PMID 28131489
- [Background] Breglia A, Godi I, Virzi GM, Guglielmetti G, Iannucci G, De Cal M, Brocca A, Carta M, Giavarina D, Ankawi G, Passannante A, Yun X, Biolo G, Ronco C. Subclinical Contrast-Induced Acute Kidney Injury in Patients Undergoing Cerebral Computed Tomography. Cardiorenal Med. 2020;10(2):125-136. doi: 10.1159/000505422. Epub 2020 Feb 7. PMID 32036364
- [Background] Suva M, Kala P, Poloczek M, Kanovsky J, Stipal R, Radvan M, Hlasensky J, Hudec M, Brazdil V, Rehorova J. Contrast-induced acute kidney injury and its contemporary prevention. Front Cardiovasc Med. 2022 Dec 6;9:1073072. doi: 10.3389/fcvm.2022.1073072. eCollection 2022. PMID 36561776
- See also: KDIGO Clinical Practice Guideline for Acute Kidney Injury. — https://kdigo.org/guidelines/acute-kidney-injury/
- See also: American College of Cardiology resources on acute coronary syndromes and PCI. — https://www.acc.org/latest-in-cardiology
- See also: SPIRIT recommendations for protocol design and structure. — https://www.spirit-statement.org
- See also: CONSORT guidelines for clinical trial reporting. — https://www.consort-statement.org/